CLINICAL TRIAL: NCT02951624
Title: The Effect of Frequency and Duration of Breaks in Sitting Time on Metabolic Cardiovascular Risk Factors
Acronym: BPS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mathias Ried-Larsen, Group leader, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 53476
Record Dates: First submitted 2016-10-30; First posted 2016-11-01 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Sedentary Lifestyle; Overweight and Obesity; Metabolic Disease
Keywords: Exercise; Breaking prolonged sitting; physical activity
MeSH Terms: conditions — Sedentary Behavior; Overweight; Obesity; Metabolic Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Experimental): Participants will spend 8 hours sedentary. Sedentary time will be spent sitting in a chair, restricted to sedentary behaviors (working on a computer, reading, watching TV, etc.) Participants will only be allowed to stand or walk to go to the toilet.
  Interventions: Behavioral: Control
- Breaker (Experimental): Participants will spend a total of 7 hours and 12 min sedentary and a total of 48 min breaking sitting time with LPA. Sedentary time will be done in bouts of 18 min with 2 min of light walking.
  Interventions: Behavioral: Breaker
- Intermediate (Experimental): Total duration of sedentary time and LPA time will be the same as in Breaker. Sedentary time will be done in bouts of 54 min with 6 min of LPA between each bout.
  Interventions: Behavioral: Intermediate
- Prolonger (Experimental): Total duration of sedentary time and LPA time will be the same as in Breaker. Sedentary time will be done in bouts of 108 min with 12 min of LPA between each bout.
  Interventions: Behavioral: Prolonger

INTERVENTIONS:
Behavioral: Control — Control intervention
  Arms: Control
Behavioral: Breaker — Short breaks of physical activity
  Arms: Breaker
Behavioral: Prolonger — longer breaks of physical activity
  Arms: Prolonger
Behavioral: Intermediate — Intermediate breaks of physical activity
  Arms: Intermediate

SUMMARY:
The primary aim of this study is to investigate the acute effect of the frequency and duration of breaks in sitting time on the metabolic risk factor profile.

DETAILED DESCRIPTION:
Fifteen (n=15) sedentary adult overweight males will be included in the study. All participants will undergo the four interventions in a randomized cross-over design. Wash out between intervention will be minimum four days.

Control (CON): Participants will be sedentary. Sedentary time will be spent sitting in a chair, restricted to sedentary behaviors (working on a computer, reading, watching TV, etc.), with a target MET below 1.5 (i.e. 1.5 times REE). Participants will only be allowed to stand or walk to go to the toilet.

Breaker: Participants will be breaking up prolonged sitting with 2 min intervals of low intensity walking.

Intermediate: Participants will be breaking up prolonged sitting with 6 min intervals of low intensity walking

Prolonger: Participants will be breaking up prolonged sitting with 12 min intervals of low intensity walking

All interventions will be matched for total physical activity as well as sitting. Thus, we aim for the active interventions to be iso-caloric.

ELIGIBILITY:
Inclusion Criteria:

* Males, age 20-50 years, waist-to-height ratio ≥ 0.5 and/or waist circumference ≥ 102 cm.

Exclusion Criteria:

* Clinically diagnosed diabetes, uncontrolled hypertension, use of glucose- and/or lipid-lowering medication, smoking, evidence of thyroid, liver, lung, heart or kidney disease, non-sedentary occupation, and VO2max levels above the considered average fitness according to age (Shvartz & Reibold 1990), contraindications to increased levels of physical activity.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11; Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
AUC post prandial glucose concentration | 6 hours

SECONDARY OUTCOMES:
AUC post prandial insulin concentration | 6 hours
AUC post prandial c-peptide concentration | 6 hours
AUC post prandial triglyceride concentration | 6 hours
AUC post prandial total cholesterol concentration | 6 hours
AUC post prandial ldl concentration | 6 hours
AUC post prandial hdl concentration | 6 hours
AUC post prandial glucagon concentration | 6 hours
Mean 24 hour glucose concentration | 24 hours
Variation in 24 hour glucose concentration | 24 hours
Maximum in 24 hour glucose concentration | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Ried, PhD, Principal Investigator — Group leader
Locations (1):
- Center for Physical Activity Research, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data may be available after publication (fully anonymized) by contact the PI